CLINICAL TRIAL: NCT04506281
Title: A Randomized Controlled, Multicenter, Open-label, Phase II Clinical Study of PD1 Antibody (Toripalimab) Combined With GEMOX Chemotherapy and Lenvatinib Neoadjuvant Treatment for Resectable Intrahepatic Cholangiocarcinoma With High-risk Recurrence Factors
Brief Title: PD1 Antibody (Toripalimab), GEMOX and Lenvatinib Neoadjuvant Treatment for Resectable Intrahepatic Cholangiocarcinoma With High-risk Recurrence Factors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Xuhui Central Hospital, Shanghai (Other); Minhang Hospital, Fudan University (Unknown); Shanghai Jinshan Hospital (Other); Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zs-ICC-neoadjuvant
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Cholangiocarcinoma, Intrahepatic
Keywords: intrahepatic Cholangiocarcinoma; Lenvatinib; Gemox chemotherapy; Programmed cell death protein 1 antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant treatment (Experimental): 1. Gemox chemotherapy:
     Day1 Oxaliplatin 85mg/m2+ gemcitabine 1g/m2, Day 8 gemcitabine 1g/m2 Three weeks is a course of treatment, a total of 3 courses.
  2. Lenvatinib (8mg/d) for 9 weeks of continuous use.
  3. Toripalimab (240mg, once every 3 weeks), used 3 times. Evaluate the resectability of the operation within 2-4 weeks after the end of the neoadjuvant treatment course, and implement radical resection. All patients after resection use capecitabine 2500mg/m2 twice a day for 2 weeks, stopping for 1 week as a course of treatment, totaling 8 courses
  Interventions: Drug: neoadjuvant treatment
- Traditional group (No Intervention): No anti-tumor drug treatment before surgery. All patients undergoing resection use capecitabine 2500mg/m2 twice a day, stopping for 1 week as a course of treatment, totaling 8 courses.

INTERVENTIONS:
Drug: neoadjuvant treatment — PD1 antibody (Toripalimab) combined with GEMOX chemotherapy and Lenvatinib neoadjuvant treatment
  Arms: Neoadjuvant treatment

SUMMARY:
A randomized controlled, multi-center, open, phase II clinical study is designed to target patients with resectable intrahepatic cholangiocarcinoma with high-risk recurrence factors which has extremely low postoperative recurrence-free survival. In this study, we aim to compare the prognosis in intrahepatic cholangiocarcinoma between Toripalimab combined with Lenvatinib and GEMOX neoadjuvant treatment and the current clinical surgical treatment (traditional group).

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) is a malignant tumor of biliary epithelial cells that originates from the branches of the intrahepatic bile duct at the second level and above. Its incidence accounts for about 15%-20% of primary liver malignancies, showing a gradually increasing trend. Surgical resection is currently the main method for the treatment of ICC. The data of a large number of ICC cases show that even radical resection (R0) patients have an average survival of only 18.3 months, while for palliative resection patients, the average survival is only 6.6 months, and laparotomy patients only 5.6 months. Retrospective studies reported that positive resection margins, lymph node metastasis, lymphatic vessel invasion, nerve bundle invasion, preoperative CA199>200U/ml, multiple tumor nodules, and differentiation are the main factors affecting the survival of ICC patients after surgery. How to improve the surgical results of ICC patients, especially those with high-risk factors for postoperative recurrence, is an important way to improve the overall survival of ICC. Neoadjuvant therapy refers to some treatments taken before surgery for newly treated tumor patients who have not found distant metastasis, including chemotherapy, radiotherapy, targeted therapy, etc., to reduce tumors, reduce tumor stages, and reduce postoperative recurrence rate, prolonging survival time. Our previous study using Toripalimab combined with Lenvatinib and Gemox chemotherapy in the first-line treatment of unresectable advanced cholangiocarcinoma (NCT03951597,2020ESMO) showed that the ORR was 80% and the DCR reached 93.3%, of which 1 case was CR, 23 cases were PR, and 2 cases were successfully treated with radical resection after downstage. And the adverse reactions are controllable. These data suggest that Toripalimab combined with Lenvatinib and Gemox chemotherapy may be an ideal neoadjuvant treatment for patients with resectable intrahepatic cholangiocarcinoma with high-risk recurrence factors, needing more investigation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Sign written informed consent 2) Male or female patients aged 18-70; 3) ECOG score 0 points, Child-Pugh rating A; 4) Clinically diagnosed as ICC as a potential entry, the neoadjuvant group must be histopathologically diagnosed as intrahepatic cholangiocarcinoma before neoadjuvant, and the traditional group must be pathologically confirmed as intrahepatic cholangiocarcinoma after surgery; 5) Resectable ICC patients with high risk factors for recurrence (tumor diameter>5cm or imaging vascular invasion, multiple tumor nodules or hilar lymph node metastasis or preoperative CA199>200U/ml); 6) The functional indicators of important organs meet the following requirements

  1. Neutrophils≥1.5*109/L; platelets≥90*109/L; hemoglobin≥9g/dl; serum albumin≥3.5g/dl;
  2. Coagulation function: International standardization (prothrombin time) ratio (INR) <1.2;
  3. T3 and T4 do not exceed the normal upper and lower limits by 2 times;
  4. Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal;
  5. Serum creatinine ≤ 1.5 times the upper limit of normal, creatinine clearance ≥ 60ml/min; 7) The subject has at least 1 measurable liver disease (according to RECIST1.1); 8) For women who are not breastfeeding or pregnant, use contraception during treatment or 3 months after the end of treatment.

Exclusion Criteria:

* 1) Pathological diagnosis of hepatocellular carcinoma, mixed hepatocellular carcinoma and other non-biliary cell carcinoma malignant tumor components; 2) Patients who relapse after surgery, have received PD1 antibody, PDL1 antibody or CTLA4 antibody, lenvatinib, chemotherapy in the past; participated in other clinical trials 30 days before screening; 3) Past or simultaneous suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary carcinoma; 4) Active tuberculosis infection. Patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, no formal anti-tuberculosis treatment or tuberculosis is still active; 5) Suffer from active, known or suspected autoimmune diseases. Subjects with hypothyroidism who only need hormone replacement therapy and skin diseases without systemic therapy can be selected; 6) Past interstitial lung disease, or (non-infectious) pneumonia and need oral or intravenous steroid therapy; 7) Long-term use of systemic hormones (dose equivalent to >10mg prednisone/day) or any other form of immunosuppressive therapy is required. Subjects using inhaled or topical corticosteroids can be selected; 8) Active infections that require systemic treatment; 9) Human immunodeficiency virus (HIV, HIV1/2 antibody) positive; 10) A history of psychotropic drug abuse, alcohol or drug abuse; 11) Significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment; 12) Suspected of being allergic to study drugs; 13) Suffer from hypertension, and cannot be well controlled by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg); 14) After antiviral therapy, HBvDNA>104 copies/ml, HCV RNA>1000; 15) Accompanied by ascites, hepatic encephalopathy, Gilbert syndrome, sclerosing cholangitis, etc. Combined with insufficiency of other organs, it is expected that they cannot accept general anesthesia or hepatectomy; 16) Other factors judged by the investigator that may affect the safety of the subject or the compliance of the trial. Such as serious illnesses (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-08-10 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 18 months
  From randomization to the occurrence of the following events: disease progression prevents radical surgery; local or distant recurrence; second primary tumor; death due to various causes.

SECONDARY OUTCOMES:
Overall survival | 24 months
  the time period from the randomization of the patient to the death event due to any reason
Objective response rate | 6 months
  The proportion of patients whose tumor volume has decreased to a predetermined value
Pathological remission rate | 6 months
  the ratio of the estimated active tumor size divided by the tumor bed size
Adverse events | 12 months
  the severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD & PhD, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaib Y, El-Serag HB. The epidemiology of cholangiocarcinoma. Semin Liver Dis. 2004 May;24(2):115-25. doi: 10.1055/s-2004-828889. PMID 15192785
- [Result] Shen WF, Zhong W, Xu F, Kan T, Geng L, Xie F, Sui CJ, Yang JM. Clinicopathological and prognostic analysis of 429 patients with intrahepatic cholangiocarcinoma. World J Gastroenterol. 2009 Dec 21;15(47):5976-82. doi: 10.3748/wjg.15.5976. PMID 20014463
- [Result] Cho SY, Park SJ, Kim SH, Han SS, Kim YK, Lee KW, Lee SA, Hong EK, Lee WJ, Woo SM. Survival analysis of intrahepatic cholangiocarcinoma after resection. Ann Surg Oncol. 2010 Jul;17(7):1823-30. doi: 10.1245/s10434-010-0938-y. Epub 2010 Feb 18. PMID 20165987
- [Result] Fisher SB, Patel SH, Kooby DA, Weber S, Bloomston M, Cho C, Hatzaras I, Schmidt C, Winslow E, Staley CA 3rd, Maithel SK. Lymphovascular and perineural invasion as selection criteria for adjuvant therapy in intrahepatic cholangiocarcinoma: a multi-institution analysis. HPB (Oxford). 2012 Aug;14(8):514-22. doi: 10.1111/j.1477-2574.2012.00489.x. Epub 2012 May 22. PMID 22762399
- [Result] Yamashita Y, Taketomi A, Morita K, Fukuhara T, Ueda S, Sanefuji K, Iguchi T, Kayashima H, Sugimachi K, Maehara Y. The impact of surgical treatment and poor prognostic factors for patients with intrahepatic cholangiocarcinoma: retrospective analysis of 60 patients. Anticancer Res. 2008 Jul-Aug;28(4C):2353-9. PMID 18751418